CLINICAL TRIAL: NCT00667433
Title: CID 0706 - Safety, Tolerability, Pharmacokinetic, and Metabolic Features of Raltegravir Among African-American Men and Women With HIV Infection
Brief Title: Raltegravir as Early Therapy in African-Americans Living With HIV Study
Acronym: REAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David A Wohl, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, David A Wohl, MD, Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID 0706
Record Dates: First submitted 2008-04-22; First posted 2008-04-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: HIV; African American; treatment naïve
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm where subjects will receive Raltegravir 400 mg BID along with Truvada once a day for 104 weeks
  Interventions: Drug: Raltegravir + Truvada

INTERVENTIONS:
Drug: Raltegravir + Truvada — Raltegravir 400 mg tablet BID PO X 104 weeks; Truvada 200/300 mg tablet once a day PO x 104 weeks
  Other Names: MK-0518; Isentress; emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg

SUMMARY:
This is a single arm, longitudinal study to examine the safety, tolerability, and pharmacokinetic and metabolic characteristics of Raltegravir among 40 African-American, HIV-infected, patients.

DETAILED DESCRIPTION:
Purpose: This study will be a single arm, prospective cohort study to examine the safety, efficacy, and pharmacokinetic and metabolic characteristics of Raltegravir in African-American men and women.

Participants: 40 HIV positive, ARV treatment-naive, African-American women and men (estimated to be 70% men, 30% women)

Procedures (methods): Subjects will receive Raltegravir 400 mg BID along with Truvada for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by HIV serology or detectable viral load
* Self-described as African-American
* Less than 7 days cumulative of prior HIV therapy
* Plasma HIV RNA PCR equal to or greater than 1000 copies/mL within 90 days prior to study entry
* Able to provide informed consent
* In the opinion of the investigator, able to comply with study medication and procedures
* ALT (SGPT) < or equal to 3.0 x ULN within 45 days prior to study entry
* GRF > 59 as calculated by MDRD within 45 days prior to study entry
* All women of reproductive potential (who have not reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) must have a negative serum or urine β-HCG pregnancy test performed within 48 hours before entry.

All study volunteers must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) and, if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use at least one reliable method of contraception (e.g., condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; or hormonal-based contraception), simultaneously while receiving the protocol-specified medication(s) and for 6 weeks after stopping the medication(s). If oral birth control pills, hormone patches, or hormone injections are used for contraception, then a second method of contraception must be used.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Prior receipt of Raltegravir
* Any condition which in the opinion of the investigator is likely to interfere with follow-up or ability to take the study medication appropriately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assess Raltegravir tolerability, acceptability, and adherence among African-American men and women initiating HIV therapy. 2. Determine the pharmacokinetics of Raltegravir in African-American men and women. | 2 years

SECONDARY OUTCOMES:
Determine the pharmacokinetics of Raltegravir in African-American men and women. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David A Wohl, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Gilde LR, Wan H, Miller MD, Wenning LA, Teppler H; Protocol 004 Part II Study Team. Rapid and durable antiretroviral effect of the HIV-1 Integrase inhibitor raltegravir as part of combination therapy in treatment-naive patients with HIV-1 infection: results of a 48-week controlled study. J Acquir Immune Defic Syndr. 2007 Oct 1;46(2):125-33. doi: 10.1097/QAI.0b013e318157131c. PMID 17721395